CLINICAL TRIAL: NCT03453073
Title: Chocolate Intake and Heart Disease and Stroke in the Women's Health Initiative: a Prospective Analysis
Brief Title: Chocolate and CVD Risk in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Brooklyn College of the City University of New York (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Greenberg, Associate Professor, Brooklyn College of the City University of New York
Other Study IDs: 438347-3
Record Dates: First submitted 2018-02-18; First posted 2018-03-05 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Disease; Heart Disease; Stroke
Keywords: Coronary heart disease; stroke; chocolate consumption; postmenopausal women; nutrition; dietary intake; epidemiology
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Stroke; Coronary Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- chocolate consumption level referent: women who ate 1 oz. (28.35 g) of chocolate <1 time/month
  Interventions: Behavioral: chocolate consumption level
- chocolate consumption level 2: women who ate 1 oz. (28.35 g) of chocolate between 1 and <1.5 times/month
  Interventions: Behavioral: chocolate consumption level
- chocolate consumption level 3: women who ate 1 oz. (28.35 g) of chocolate between 1.5 and <3.5 times/month,
  Interventions: Behavioral: chocolate consumption level
- chocolate consumption level 4: women who ate 1 oz. (28.35 g) of chocolate between 3.5 times/month and <3 times/week
  Interventions: Behavioral: chocolate consumption level
- chocolate consumption level 5: women who ate 1 oz. (28.35 g) of chocolate >3 times/week
  Interventions: Behavioral: chocolate consumption level
- No physician diagnosis: No incidence of serious chronic disease prior to visit 3
  Interventions: Other: physician diagnosis of first occurrence of serious chronic disease
- Physician diagnosis: Incidence of serious chronic disease prior to visit 3
  Interventions: Other: physician diagnosis of first occurrence of serious chronic disease
- Younger: Age<65 years at follow-up baseline
  Interventions: Behavioral: chocolate consumption level
- Older: Age>=65 years at follow-up baseline
  Interventions: Behavioral: chocolate consumption level

INTERVENTIONS:
Behavioral: chocolate consumption level — level of consumption of 1 oz. of chocolate, as assessed at baseline
  Groups: Older; Younger; chocolate consumption level 2; chocolate consumption level 3; chocolate consumption level 4; chocolate consumption level 5; chocolate consumption level referent
Other: physician diagnosis of first occurrence of serious chronic disease
  Groups: No physician diagnosis; Physician diagnosis

SUMMARY:
The investigators will conduct an epidemiological analysis of data from the Women's Health Initiative to investigate the prospective association between chocolate intake and the risk of heart disease and stroke.

DETAILED DESCRIPTION:
BACKGROUND: Three recent meta-analyses found significant prospective inverse associations between chocolate intake and cardiovascular disease risk. Evidence from these meta-analyses suggests that such inverse associations may only apply to elderly individuals or those with preexisting major chronic disease.

OBJECTIVE: The investigators will assess the association between habitual chocolate intake and subsequent incident coronary heart disease (CHD) and stroke, and the potential effect of modification by age.

DESIGN: The investigators will conduct multivariable Cox regression analyses using data from 83,310 postmenopausal women free of baseline preexisting major chronic disease in the prospective Women's Health Initiative cohort. Chocolate intake was assessed using a food frequency questionnaire. Physician adjudicated events or deaths were ascertained up to September 30, 2013.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women
2. age between 50 and 79 years
3. enrolled in the Women's Health Initiative (WHI) Observational Study, or in the control arm of one or more overlapping WHI clinical trials.

Exclusion Criteria:

1. implausible energy intakes, defined as <600 kcal/d or >5,000 kcal/d;
2. implausible body mass indices (BMI) (<15 or >50 kg/m2)
3. implausible height<122 cm (4 ft.)
4. self-reported preexisting serious chronic disease at baseline, including diabetes, angina, myocardial infarction (MI), stroke, heart failure, coronary artery bypass graft, percutaneous coronary intervention or cancer.
5. missing data on preexisting major chronic disease or any exposure, outcome or confounder variables.

Ages: 55 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women 50-79 years of age
Study Population: community residents
Sampling Method: Non-Probability Sample
Enrollment: 83310 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
incidence of heart disease | between the baseline survey (1993-8) & September 30, 2013, average 13.4 years
  physician adjudicated first occurrence of, or death due to, heart disease
incidence of stroke | between the baseline survey (1993-8) & September 30, 2013, average 13.4 years
  physician adjudicated first occurrence of, or death due to, stroke
incidence of heart disease or stroke | between the baseline survey (1993-8) & September 30, 2013, average 13.4 years
  physician adjudicated first occurrence of, or death due to, heart disease or stroke
change in chocolate intake | time between the baseline and visit 3, average 3 years
  change in chocolate intake between visit 1 and 3
change in dietary energy intake | time between the baseline and year 3, average 3 years
  change in dietary energy intake between visit 1 and 3
change in dietary fat intake | time between the baseline and year 3, average 3 years
  change in dietary fat intake between visit 1 and 3
change in BMI | time between the baseline and year 3, average 3 years
  change in BMI between visit 1 and 3

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greenberg JA, Manson JE, Neuhouser ML, Tinker L, Eaton C, Johnson KC, Shikany JM. Chocolate intake and heart disease and stroke in the Women's Health Initiative: a prospective analysis. Am J Clin Nutr. 2018 Jul 1;108(1):41-48. doi: 10.1093/ajcn/nqy073. PMID 29931040